CLINICAL TRIAL: NCT01508806
Title: A Single-centre, Open-label, Trial Investigating the Pharmacokinetics and the Tolerability of Liraglutide in Subjects With Normal Renal Function and in Subjects With Impaired Renal Function
Brief Title: Safety and Tolerability of Liraglutide in Subjects With Impaired Kidney Function and in Subjects With Normal Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-1329
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Normal renal function (Experimental)
  Interventions: Drug: liraglutide
- Mild renal impairment (Experimental)
  Interventions: Drug: liraglutide
- Moderate renal impairment (Experimental)
  Interventions: Drug: liraglutide
- Severe renal impairment (Experimental)
  Interventions: Drug: liraglutide
- End-stage renal disease (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Single dose of 0.75 mg, administered as a subcutaneous injection

SUMMARY:
This trial is conducted in Oceania. The aim of this trial is to assess whether dose adjustment is required for patients with renal impairment by investigating the pharmacokinetics of liraglutide in subjects with various degrees of renal impairment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting the pre-defined GFR (glomerular filtration rate) criteria (estimated by the Cockcroft and Gault formula) for any of the renal function groups
* Body Mass Index (BMI) maximum 40 kg/m^2

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products
* Renal transplanted patients
* Haemodialysis patients
* Cardiac problems
* Uncontrolled treated/untreated hypertension
* History of alcoholism or drug abuse during the last 12 months
* Smoking of more than 10 cigarettes per day, or the equivalent for other tobacco products
* Habitual excessive consumption of methylxanthine-containing beverages and foods (coffee, tea, soft drinks such as cola, chocolate) as judged by the investigator
* Excessive consumption of food deviating from a normal diet as judged by the Investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-08; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Area under the Curve (AUC)

SECONDARY OUTCOMES:
AUC (0-t)
Cmax, maximum concentration
tmax, time to reach Cmax
t½, terminal half-life
CLR (renal clearance)
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Christchurch, Australia

REFERENCES:
- [Result] Jacobsen LV, Hindsberger C, Robson R, Zdravkovic M. Effect of renal impairment on the pharmacokinetics of the GLP-1 analogue liraglutide. Br J Clin Pharmacol. 2009 Dec;68(6):898-905. doi: 10.1111/j.1365-2125.2009.03536.x. PMID 20002084
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com